CLINICAL TRIAL: NCT00317109
Title: Booster Vaccination Study to Assess Safety & Reactogenicity of a Dose of DTPw-HBV/Hib Vaccine and to Assess the Immunogenicity, Safety & Reactogenicity of a Dose of Mencevax™ ACW in Subjects Primed in Study 759346/007
Brief Title: Study to Asses DTPw-HBV/Hib at 15-18 Months (m) and Mencevax™ ACW at 24 to 30 m in Primed Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104756
Record Dates: First submitted 2006-02-03; First posted 2006-04-24 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-01

CONDITIONS: Infections, Meningococcal
Keywords: meningococcal serogroups A and C diseases; tetanus; hepatitis B; pertussis; Haemophilus influenzae type b; meningococcal vaccine; Prophylaxis diphtheria
MeSH Terms: conditions — Meningococcal Infections; Tetanus; Hepatitis B; Whooping Cough; Haemophilus Infections | interventions — Hiberix

ARMS (2):
- AC primed Group (Experimental)
  Interventions: Biological: Tritanrix™- HepB; Biological: Hiberix™; Biological: Mencevax™ ACW
- AC unprimed Group (Active Comparator)
  Interventions: Biological: Tritanrix™- HepB; Biological: Hiberix™; Biological: Mencevax™ ACW

INTERVENTIONS:
Biological: Tritanrix™- HepB — One intramuscular dose during the booster vaccination study in subjects aged 15 to 18 months
Biological: Hiberix™ — One intramuscular dose during the booster vaccination study in subjects aged 15 to 18 months
Biological: Mencevax™ ACW — One subcutaneous dose during the booster vaccination study in subjects aged 24 to 30 months

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of a booster dose of diphtheria-tetanus-whole cell pertussis-hepatitis B virus/Haemophilus influenzae type b vaccine (DTPw-HBV/Hib) at 15-18 m and to assess the immunogenicity, safety, and reactogenicity of a dose of Mencevax™ Group A, C and W135 polysaccharide meningococcal vaccine (ACW) at 24 to 30 m in primed subjects.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This open study will have two parallel groups based on the vaccination received in the primary study: AC primed Group: primed with Tritanrix™-HepB/Hib-MenAC vaccine and AC unprimed Group (control): primed with Tritanrix™-HepB/Hiberix™ vaccine. All subjects will receive a booster dose of Tritanrix™-HepB/Hiberix™ vaccine at 15 to 18 months of age with GSK Biological's OPV vaccine given concomitantly and a dose of Mencevax™ ACW vaccine at 24 to 30 months of age. Blood sampling will be done prior to (pre) and one month after (post) the Mencevax™ ACW vaccine administration for immunogenicity analyses. The study will last minimum 7 to maximum 16 months per subject.

Mencevax™ ACWY was changed to Mencevax™ ACW throughout the posting to correct an inconsistency in the earlier version of the protocol posting and to reflect the actual situation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 15 and 18 months of age at the time of vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having participated in the primary vaccination study (CPMS N° 759346/007).

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the vaccination, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of vaccination.
* Booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib) and/or meningococcal serogroups A, C or W disease, after the date of the study conclusion visit of the primary vaccination study (CPMS N° 759346/007).
* History of diphtheria, tetanus, pertussis, hepatitis B, Hib and/or meningococcal serogroup A, C or W disease.
* Known exposure to diphtheria, tetanus, pertussis, hepatitis B, Hib and/or meningococcal serogroup A, C or W disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines administered in the study.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures including febrile seizures in infancy.
* Acute disease at the time of enrolment.
* Axillary temperature ≥ 37.5°C at the time of vaccination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the vaccination or planned administration during the study period.
* Anaphylactic reaction following the administration of vaccine in the primary vaccination study.
* Known hypersensitivity to any component of the vaccine, or subjects having shown signs of hypersensitivity after previous administration of diphtheria, tetanus, pertussis, hepatitis B, Hib or meningococcal vaccines.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2006-04-19; Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- South Africa (3):
  - GSK Investigational Site, Brits
  - GSK Investigational Site, Ga-Rankuwa
  - GSK Investigational Site, Rooihuiskraal

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tritanrix-HepB/Hiberix Group: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317122), were boosted in the current study with one dose of the same vaccine at 15 to 18 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACW vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
- Tritanrix-HepB/Hiberix-Mencevax AC Group: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix-Mencevax AC vaccine in the primary study (NCT00317122), were boosted in the current study with one dose of Tritanrix-HepB/Hiberix vaccine at 15 to 18 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACW vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
Period: Overall Study
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Started | 84 | 84
Completed | 81 | 84
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Migated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Months at TRITANRIX™-HEPB/HIBERIX™ booster | 16.5 (1.02) | 16.5 (1.02) | 16.5 (1.02)
  Months at MENCEVAX™ booster | 24.5 (0.92) | 24.6 (1.04) | 24.55 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 84
  Male | 39 | 45 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Against N. Meningitidis Serogroups A, C Using Rabbit Complement (rSBA-MenA,C) Antibodies
Description: Pre-defined assay cut-off values for assessed titers were greater than or equal to (≥) 1:128.
Time Frame: At one month post vaccination with Mencevax™ ACW vaccine (Month 25-31)
Population: The analysis were performed on the Booster ATP cohort for immunogenicity which included all evaluable subjects who received the 3 vaccine doses in the primary vaccination study, received one of the two vaccines according to the protocol in this booster study and for whom data concerning immunogenicity measures were available.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 65 | 66
Subjects
  rSBA-MenA [N=65,60] | 65 | 59
  rSBA-MenC [N=59,66] | 30 | 66

2. Secondary Outcome: Number of Subjects With rSBA-MenA,C, W-135 Antibody Titers ≥ Predefined Cut-offs
Description: Antibody titer cut-offs were ≥ 1:8 and ≥ 1:128.
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 67 | 66
Subjects
  rSBA-MenA ≥1:8 (M24-30) [N=58,53] | 55 | 50
  rSBA-MenA ≥1:8 (M25-31) [N=65,60] | 65 | 60
  rSBA-MenA ≥1:128 (M24-30) [N=58,53] | 54 | 48
  rSBA-MenC ≥1:8 (M24-30) [N=67,61] | 10 | 42
  rSBA-MenC ≥1:8 (M25-31) [N=59,66] | 53 | 66
  rSBA-MenC ≥1:128 (M24-30) [N=67,61] | 4 | 27
  rSBA-MenW-135 ≥1:8 (M24-30) [N=67,63] | 18 | 20
  rSBA-MenW-135 ≥1:8 (M25-31) [N=64,66] | 49 | 44
  rSBA-MenW-135 ≥1:128 (M24-30) [N=67,63] | 13 | 11
  rSBA-MenW-135 ≥1:128 (M25-31) [N=64,66] | 45 | 37

3. Secondary Outcome: Anti-rSBA-MenA, C, W-135 Antibody Titers
Description: Antibody titers were expressed as geometric mean titers (GMTs).
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 67 | 66
Titers
  rSBA-MenA (M24-30) [N=58,53] | 503.8 [346.6 to 732.1] | 509.9 [326.9 to 795.3]
  rSBA-MenA (M25-31) [N=65,60] | 1871.7 [1515.2 to 2311.9] | 1562.0 [1252.9 to 1947.2]
  rSBA-MenC (M24-30) [N=67,61] | 6.7 [4.9 to 9.1] | 50.7 [30.7 to 83.5]
  rSBA-MenC (M25-31) [N=59,66] | 141.3 [89.2 to 223.9] | 5251.6 [3662.5 to 7530.2]
  rSBA-MenW-135 (M24-30) [N=67,63] | 11.1 [7.2 to 17.1] | 13.7 [8.3 to 22.5]
  rSBA-MenW-135 (M25-31) [N=64,66] | 159.4 [91.5 to 277.6] | 92.8 [50.6 to 170.0]

4. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA) and C (Anti-PSC) Antibody Concentrations Above Predefined Cut-off Values
Description: Antibody concentrations cut-off were ≥ 0.3 and ≥2 micrograms per millilitre (µg/mL).
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 65 | 66
Subjects
  anti-PSA ≥ 0.3 µg/mL (M24-30) [N=63,61] | 8 | 10
  anti-PSA ≥ 0.3 µg/mL (M25-31) [N=65,65] | 62 | 64
  anti-PSA ≥ 2 µg/mL (M24-30) [N=63,61] | 0 | 1
  anti-PSA ≥ 2 µg/mL (M25-31) [N=65,65] | 48 | 64
  anti-PSC ≥ 0.3 µg/mL (M24-30) [N=61,64] | 6 | 33
  anti-PSC ≥ 0.3 µg/mL (M25-31) [N=65,66] | 65 | 66
  anti-PSC ≥ 2 µg/mL (M24-30) [N=61,64] | 2 | 4
  anti-PSC ≥ 2 µg/mL (M25-31) [N=65,66] | 64 | 65

5. Secondary Outcome: Anti-PSA and Anti-PSC Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 65 | 66
µg/mL
  anti-PSA (M24-30) [N=63,61] | 0.18 [0.16 to 0.20] | 0.19 [0.16 to 0.21]
  anti-PSA (M25-31) [N=65,65] | 6.61 [4.27 to 10.22] | 22.39 [16.11 to 31.10]
  anti-PSC (M24-30) [N=61,64] | 0.18 [0.15 to 0.22] | 0.35 [0.27 to 0.44]
  anti-PSC (M25-31) [N=65,66] | 15.70 [12.54 to 19.65] | 35.10 [27.40 to 44.96]

6. Secondary Outcome: Number of Subjects With Anti- Polysaccharide W (Anti-PSW) Antibody Concentrations ≥ Predefined Cut-off Values
Description: Antibody concentrations were ≥ 0.3 µg/mL.
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 64 | 66
Subjects
  anti-PSW (M24-30) [N=61,62] | 0 | 2
  anti-PSW (M25-31) [N=64,66] | 64 | 64

7. Secondary Outcome: Anti-PSW Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to (Months 24-30) & one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 64 | 66
µg/mL
  anti-PSW (M24-30) [N=61,62] | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.18]
  anti-PSW (M25-31) [N=64,66] | 4.89 [3.68 to 6.50] | 5.19 [3.63 to 7.40]

8. Secondary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentrations ≥ Predefined Cut-off Values
Description: Antibody concentrations cut-off were ≥ 10 milli international units per milliliter (mIU/mL).
Time Frame: Prior to (Months 24-30) the administration of the Mencevax™ ACW vaccine
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 66 | 66
Subjects | 63 | 65

9. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to (Months 24-30) the administration of the Mencevax™ ACW vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 66 | 66
mIU/mL | 722.0 [456.2 to 1142.8] | 713.1 [438.2 to 1160.5]

10. Secondary Outcome: Number of Subjects With Vaccine Response for rSBA-Men A, C and W-135
Description: Vaccine response was defined as follows: for initially seronegative subjects (i.e. with rSBA titre < 1:8 pre-vaccination), rSBA titre ≥ 1:32 post-vaccination (seroconversion), and for initially seropositive subjects (i.e. with rSBA titre ≥ 1:8 pre-vaccination), at least a 4-fold increase in rSBA titre from pre to post-vaccination.
Time Frame: At one month after the administration of the Mencevax™ ACW vaccine (Months 25-31)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 64 | 62
Subjects
  rSBA-MenA, Total [N=56,47] | 26 | 21
  rSBA-MenC, Total [N=59,60] | 41 | 56
  rSBA-MenW-135, Total [N=64,62] | 41 | 32

11. Secondary Outcome: Number of Subjects With Fever
Description: Any Fever (measured rectally) = subjects with symptom, regardless of the intensity grade.
Time Frame: During the 4-day (Days 0-3) after the administration of the Tritanrix™-HepB/Hiberix™ vaccine
Population: The analysis was performed on the Booster Total Vaccinated Cohort which included all subjects who received at least one of the two vaccines.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 84 | 84
Subjects | 33 | 29

12. Secondary Outcome: Number of Subjects With Solicited Local Symtoms
Description: Assessed solicited local symptoms were: pain, redness and swelling at the injection site. Any = subjects with symptom, regardless of the intensity grade.
Time Frame: During the 4-Day (Days 0-3) after the administration of the Mencevax™ ACW vaccine
Population: The analysis was performed on the Booster Total Vaccinated Cohort which included all subjects who received at least one of the two vaccines and had the symptoms sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 80 | 82
Subjects
  Any Pain | 21 | 25
  Any Redness | 20 | 16
  Any Swelling | 13 | 11

13. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were: drowsiness, fever, irritability and loss of appetite. Any = subjects with symptoms, regardless of intensity grade and casual relationship to study vaccination.
Time Frame: During the 4-Day (Days 0-3) after the administration of the Mencevax™ ACW vaccine
Population: The analysis were performed on the Booster Total Vaccinated Cohort which included all subjects who received at least one of the two vaccines and had the symptoms sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 80 | 83
Subjects
  Any Drowsiness | 14 | 12
  Any Fever | 8 | 5
  Any Irritability | 15 | 12
  Any Loss of appetite | 13 | 18

14. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-Day (Days 0-30) after the administration of the Mencevax™ ACW vaccine
Population: The analysis were performed on the Booster Total Vaccinated Cohort which included all subjects who received at least one of the two vaccines.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 82 | 84
Subjects | 10 | 16

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Months 15-18 and up to Months 25-31 post vaccination
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Number analyzed (Participants) | 82 | 84
Subjects | 2 | 1

ADVERSE EVENTS:
Time Frame: Fever during the 4-day (Days 0-3) post Tritanrix-HepB/Hiberix vaccination; Solicited local/general during the 4-day (Days 0-3) and AEs during the 31-day (Days 0-30) after Mencevax ACW vaccination; SAEs from Months 15-18 and up to Months 25-31.
Arm/Group | Tritanrix-HepB/Hiberix Group | Tritanrix-HepB/Hiberix-Mencevax AC Group
Serious Adverse Events (participants affected / at risk) | 2/82 | 1/84
Other Adverse Events (participants affected / at risk) | 56/84 | 56/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tritanrix-HepB/Hiberix Group (N=82) | Tritanrix-HepB/Hiberix-Mencevax AC Group (N=84)
Febrile convulsion (Nervous system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tritanrix-HepB/Hiberix Group (N=84) | Tritanrix-HepB/Hiberix-Mencevax AC Group (N=84)
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Pain (General disorders) | 21 | 25/82
Redness (General disorders) | 20 | 16/82
Swelling (General disorders) | 13 | 11/82
Drowsiness (General disorders) | 14 | 12/83
Fever/(Rectally) (°C) (General disorders) | 8 | 5/83
Irritability (General disorders) | 15 | 12/83
Loss of appetite (General disorders) | 13 | 18/83

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.